CLINICAL TRIAL: NCT06569914
Title: Study on the Influence of Humanized Nursing Model on the Effect of Intravenous Infusion Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY-2024-141
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Intravenous Infusion
Keywords: Humanized nursing; Intravenous infusion; Psychological state score; Adverse reaction incidence rate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Routine nursing:strict implementation of the "three checks and eight pairs" process, strict inspection of the quality of drugs used by patients, and strict adherence to medical advice on drug dosage.
- observation group (Experimental): humanistic nursing：(1) Humanized environmental care；(2) Humanized medical guidance；(3)Humanized psychological nursing；(4) Humanized and standardized management of IVGTT treatment process
  Interventions: Behavioral: Humanized care

INTERVENTIONS:
Behavioral: Humanized care — (1) Humanized environmental care；(2) Humanized medical guidance；(3)Humanized psychological nursing；(4) Humanized and standardized management of IVGTT treatment process
  Arms: observation group

SUMMARY:
The routine nursing content is relatively simple, and nursing measures are greatly influenced by the personal experience of nursing staff, lacking a systematic approach Sexuality, scientificity, and relatively late implementation have resulted in unsatisfactory preventive effects. Early nursing intervention emphasizes the importance of patients The impact of early postoperative intervention can effectively meet the cognitive needs of patients and improve their compliance with treatment and care At the same time, early intervention can help patients avoid risks and better achieve nursing goals. This selection A study was conducted on 40 patients receiving intravenous infusion to explore the impact of humanized nursing on the effectiveness of intravenous infusion nursing.

DETAILED DESCRIPTION:
Forty patients who chose our hospital for intravenous infusion were included in the study. Randomly divide two groups using the numerical table method.Control group, 20 cases, receiving routine nursing care.Observation group, 20 cases, receiving humanized care.

Control group: Routine nursing, strict implementation of the "three checks and eight pairs" process, strict inspection of the quality of drugs used by patients, and strict adherence to medical advice on drug dosage.

Observation group: Humanized nursing includes humanized environmental care, humanized medical guidance, humanized psychological care, and humanized standardized management of IVGTT treatment process. The specific content is: (1) Humanized environmental care: Increase the frequency of cleaning the ward. If there is vomit or stagnant water, it should be removed as soon as possible to ensure that the ward floor is always kept clean and tidy, and to avoid patients falling due to water stains or foreign objects on the floor. Reasonably increase the number of garbage bins in the ward area. If conditions permit, place magazines, educational manuals, and other items in the ward that can help patients pass the time during the infusion process. (2) Humanized medical guidance: In addition to inquiring about the patient's allergy history and explaining the effects of medication before infusion, explain possible adverse reactions and corresponding treatment measures to the patient to avoid confusion, negative emotions or psychology after adverse reactions occur. If the patient does not have good vascular conditions, nursing staff can help massage the venous area before puncture, if the condition allows. Inform patients to pay attention to any adverse events (such as slipping of infusion set, redness and swelling of puncture site, etc.) during infusion, and immediately notify nursing staff if any are found. (3) Humanized psychological nursing: Many patients resist venipuncture, and nursing staff need to provide health education before IVGTT, so that patients understand the necessity and safety of IVGTT, improve patient cooperation, actively communicate with patients, understand their concerns about IVGTT, and provide timely and correct guidance; Remind family members to care for and encourage patients, so that they can actively cooperate with IVGTT. (4) Humanized and standardized management of IVGTT treatment process: One of the core tasks of nursing work is IVGTT. We strictly follow the hospital's nursing system for IVGTT treatment, strengthen training for nursing staff in terms of service attitude, social skills, puncture skills, etc., comprehensively improve the personal comprehensive literacy of nursing staff, and ensure that all nursing staff can perform venous puncture in a standardized and efficient manner.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving intravenous infusion in our hospital
* Have complete clinical data
* Know and sign the informed consent form

Exclusion Criteria:

* Underage patients
* Patients with consciousness and cognitive impairments
* Patients with mental illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale | Up to 24 hours (during intravenous infusion)
  Evaluate patients' psychological changes through the four indicators in the Hamilton Depression Scale (depression, mental anxiety, sleep disorders, and physical anxiety). Each indicator ranges from 0 to 4 points, with 0 being the minimum value and 4 being the maximum value. The better the patient's mentality, the lower the score.
Self-made scale | Up to 24 hours (during intravenous infusion)
  Evaluate patients' satisfaction with nursing services through five indicators in a self-made scale (environmental quality, reception attitude, puncture proficiency, health education quality, communication ability). The range of each indicator is from 0 to 100 points, with 0 being the minimum value and 100 being the maximum value. The higher the patient satisfaction, the higher the rating.

CONTACTS AND LOCATIONS:
Locations (1):
- the Fourth Affiliated Hospital of School of Medicine, and International School of Medicine, International Institutes of Medicine, Yiwu, ZhengJiang, China